CLINICAL TRIAL: NCT06524258
Title: Testicular Elastography for Predicting the Likelihood of Sperm Retrieval in Microscopic Testicular Sperm Extraction
Brief Title: Testicular Elastography for Microscopic Testicular Sperm Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: Harran University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRÜ-TUNÇEKİN-001
Record Dates: First submitted 2024-07-16; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Azoospermia; Elasticity Imaging Techniques; Fertility Preservation
Keywords: share wave elastography; microscopic testicular sperm extraction; azoospermia
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tese positive (Other): micro tese positive
  Interventions: Diagnostic Test: testicular elastography
- tese negative (Other): micro tese negative
  Interventions: Diagnostic Test: testicular elastography

INTERVENTIONS:
Diagnostic Test: testicular elastography — testicular elastography for predicting non obstructive azoospermia

SUMMARY:
Before commencing our study, we obtained approval from the local ethics committee. The study focused on patients who visited our urology outpatient clinic for infertility between January 2020 and March 2021. Eighty-four patients diagnosed with non-obstructive azoospermia were prospectively enrolled in the study.

Azoospermia was diagnosed after performing semen analysis at least twice, adhering to the criteria outlined by the WHO. All patients underwent karyotype analysis and Y microdeletion analysis. Testicular volumes were measured using Prader orchidometry and confirmed by scrotal ultrasonography.

For patients scheduled for Micro-TESE, elastography measurements were conducted in the supine position. These measurements were performed by the same radiologist in the Radiology department. A total of six points Shear Wave Elastography (SWE) measurements were recorded from each patient, including upper right, middle right, lower right, upper left, middle left, and lower left.

All patients underwent the micro-TESE procedure by the same surgeon. The procedure was first applied to the testis with a better volume and consistency. Samples of large and bright tubules were extracted using microforceps under a microscope, utilizing a magnification range of 20X-25X. The tissues obtained were subsequently assessed by the same embryologist who was present in the operating room. The embryologist provides biopsy results indicating the presence or absence of spermatozoa. If five or more mature spermatozoa are observed within the testicular tissues, the procedure is terminated. However, if fewer than five spermatozoa are identified in the tissues, the procedure is repeated on the contralateral testicle to ensure a comprehensive examination and thorough exploration. Tissues containing a satisfactory quantity of sperm were processed and preserved in the incubator until the Intracytoplasmic Sperm Injection (ICSI) procedure which was planned following the sperm cryopreservation of the patients whose sperms could be retrieved. In cases where sperm could not be retrieved from patients, testicular tissue was placed in Bouin's solution and sent for histopathological examination.

DETAILED DESCRIPTION:
Before commencing our study, we obtained approval from the local ethics committee. The study focused on patients who visited our urology outpatient clinic for infertility between January 2020 and March 2021. Eighty-four patients diagnosed with non-obstructive azoospermia were prospectively enrolled in the study. Patients with obstructive azoospermia, hypogonadotropic hypogonadism, history of previous testicular disease, previous TESE, and history of chemotherapy or radiotherapy were excluded from the study.

Azoospermia was diagnosed after performing semen analysis at least twice, adhering to the criteria outlined by the WHO. All patients underwent karyotype analysis and Y microdeletion analysis. Testicular volumes were measured using Prader orchidometry and confirmed by scrotal ultrasonography.

For patients scheduled for Micro-TESE, elastography measurements were conducted in the supine position. These measurements were performed by the same radiologist in the Radiology department. A total of six points Shear Wave Elastography (SWE) measurements were recorded from each patient, including upper right, middle right, lower right, upper left, middle left, and lower left.

All patients underwent the micro-TESE procedure by the same surgeon. The procedure was first applied to the testis with a better volume and consistency. Samples of large and bright tubules were extracted using microforceps under a microscope, utilizing a magnification range of 20X-25X. The embryologist provides biopsy results indicating the presence or absence of spermatozoa. If five or more mature spermatozoa are observed within the testicular tissues, the procedure is terminated. However, if fewer than five spermatozoa are identified in the tissues, the procedure is repeated on the contralateral testicle to ensure a comprehensive examination and thorough exploration. Tissues containing a satisfactory quantity of sperm were processed and preserved in the incubator until the Intracytoplasmic Sperm Injection (ICSI) procedure which was planned following the sperm cryopreservation of the patients whose sperms could be retrieved. In cases where sperm could not be retrieved from patients, testicular tissue was placed in Bouin's solution and sent for histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* non obstructive azoospermia
* testicular elastography performed
* micro tese performed

Exclusion Criteria:

* obstructive azoospermia
* testicular elastography not performed
* micro tese not performed

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
shear wave elastography right upper pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the right upper pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.
shear wave elastography right middle pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the right middle pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.
shear wave elastography right lower pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the right lower pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.
shear wave elastography left upper pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the left upper pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.
shear wave elastography left middle pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the left middle pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.
shear wave elastography left lower pole of the testes | 1 day before micro-TESE surgery
  Elastography measurements of the left lower pole of the testes were conducted in all patients in the supine position using ultrasonography before the operation.

SECONDARY OUTCOMES:
micro-tese surgery sperm retrieval | 1 day after shear wave elastography measurement
  All patients underwent the micro-TESE procedure by the same surgeon.Patients were evaluated as positive or negative based on sperm retrieval results.

CONTACTS AND LOCATIONS:
Overall Officials: ADEM TUNÇEKİN, Study Chair — Harran University
Locations (1):
- Harran Üniversitesi, Sanliurfa, Halilye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, Vanderpoel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) revised glossary of ART terminology, 2009. Fertil Steril. 2009 Nov;92(5):1520-4. doi: 10.1016/j.fertnstert.2009.09.009. Epub 2009 Oct 14. PMID 19828144
- [Background] Agarwal A, Baskaran S, Parekh N, Cho CL, Henkel R, Vij S, Arafa M, Panner Selvam MK, Shah R. Male infertility. Lancet. 2021 Jan 23;397(10271):319-333. doi: 10.1016/S0140-6736(20)32667-2. Epub 2020 Dec 10. PMID 33308486
- [Background] Sharlip ID, Jarow JP, Belker AM, Lipshultz LI, Sigman M, Thomas AJ, Schlegel PN, Howards SS, Nehra A, Damewood MD, Overstreet JW, Sadovsky R. Best practice policies for male infertility. Fertil Steril. 2002 May;77(5):873-82. doi: 10.1016/s0015-0282(02)03105-9. No abstract available. PMID 12009338
- [Background] Sharma M, Leslie SW. Azoospermia. 2023 Nov 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK578191/ PMID 35201719
- [Background] Practice Committee of American Society for Reproductive Medicine in collaboration with Society for Male Reproduction and Urology. The management of infertility due to obstructive azoospermia. Fertil Steril. 2008 Nov;90(5 Suppl):S121-4. doi: 10.1016/j.fertnstert.2008.08.096. PMID 19007607
- [Background] Bernie AM, Ramasamy R, Schlegel PN. Predictive factors of successful microdissection testicular sperm extraction. Basic Clin Androl. 2013 Oct 2;23:5. doi: 10.1186/2051-4190-23-5. eCollection 2013. PMID 25763186
- [Background] Flannigan R, Bach PV, Schlegel PN. Microdissection testicular sperm extraction. Transl Androl Urol. 2017 Aug;6(4):745-752. doi: 10.21037/tau.2017.07.07. PMID 28904907
- [Background] Baleato-Gonzalez S, Osorio-Vazquez I, Flores-Rios E, Santiago-Perez MI, Laguna-Reyes JP, Garcia-Figueiras R. Testicular Evaluation Using Shear Wave Elastography (SWE) in Patients with Varicocele. J Imaging. 2023 Aug 22;9(9):166. doi: 10.3390/jimaging9090166. PMID 37754930
- [Background] Schurich M, Aigner F, Frauscher F, Pallwein L. The role of ultrasound in assessment of male fertility. Eur J Obstet Gynecol Reprod Biol. 2009 May;144 Suppl 1:S192-8. doi: 10.1016/j.ejogrb.2009.02.034. Epub 2009 Mar 20. PMID 19303691
- [Background] Herek D, Cakmak V, Comut E, Herek O. The value of multimodal ultrasonography in the evaluation of late presenting testicular torsion in a rat experimental model. Br J Radiol. 2024 Feb 2;97(1154):377-385. doi: 10.1093/bjr/tqad059. PMID 38302083
- [Background] Lin YY, Mao L, Li J, Zhu ZM, Luo YH, Zhou XH, Qiu SD, Chen F. Exploring the anatomical factors influencing testes elasticity via ultrasound shear wave elastography: Preliminary results. Rev Int Androl. 2023 Oct-Dec;21(4):100367. doi: 10.1016/j.androl.2023.100367. Epub 2023 Jul 7. PMID 37422973
- [Background] Illiano E, Trama F, Ruffo A, Romeo G, Riccardo F, Crocetto F, Iacono F, Costantini E. Testicular shear wave elastography in oligo-astheno-teratozoospermic individuals: a prospective case-control study. Int Urol Nephrol. 2021 Sep;53(9):1773-1783. doi: 10.1007/s11255-021-02909-4. Epub 2021 Jun 10. PMID 34114152
- [Background] Harris SE, Sandlow JI. Sperm acquisition in nonobstructive azoospermia: what are the options? Urol Clin North Am. 2008 May;35(2):235-42, ix. doi: 10.1016/j.ucl.2008.01.008. PMID 18423244
- [Background] Schlegel PN. Testicular sperm extraction: microdissection improves sperm yield with minimal tissue excision. Hum Reprod. 1999 Jan;14(1):131-5. doi: 10.1093/humrep/14.1.131. PMID 10374109
- [Background] Arian I, Dumbraveanu I, Ghenciu V, Machidon D, Ernu I, Ceban E. Histological and immunohistochemical outcomes after microdissection TESE in contrast with hormonal profile, testis volume and genetics in patients with azoospermia. J Med Life. 2023 Jan;16(1):144-152. doi: 10.25122/jml-2022-0336. PMID 36873127
- [Background] Marcon J, Trottmann M, Rubenthaler J, D'Anastasi M, Stief CG, Reiser MF, Clevert DA. Three-dimensional vs. two-dimensional shear-wave elastography of the testes - preliminary study on a healthy collective. Clin Hemorheol Microcirc. 2016;64(3):447-456. doi: 10.3233/CH-168115. PMID 27886002
- [Background] Ozturker C, Karagoz E, Incedayi M. Non-Invasive Evaluation of Liver Fibrosis: 2-D Shear Wave Elastography, Transient Elastography or Acoustic Radiation Force Impulse Imaging? Ultrasound Med Biol. 2016 Dec;42(12):3052. doi: 10.1016/j.ultrasmedbio.2016.03.033. Epub 2016 May 17. No abstract available. PMID 27207019
- [Background] Magri F, Chytiris S, Capelli V, Alessi S, Nalon E, Rotondi M, Cassibba S, Calliada F, Chiovato L. Shear wave elastography in the diagnosis of thyroid nodules: feasibility in the case of coexistent chronic autoimmune Hashimoto's thyroiditis. Clin Endocrinol (Oxf). 2012 Jan;76(1):137-41. doi: 10.1111/j.1365-2265.2011.04170.x. PMID 21740455
- [Background] Marsaud A, Durand M, Raffaelli C, Carpentier X, Rouscoff Y, Tibi B, Floc'h A, De Villeneuve MH, Haider R, Ambrosetti D, Fontas E, Padovani B, Amiel J, Chevallier D. [Elastography shows promise in testicular cancer detection]. Prog Urol. 2015 Feb;25(2):75-82. doi: 10.1016/j.purol.2014.11.008. Epub 2014 Dec 30. French. PMID 25555503
- [Background] Zhang X, Lv F, Tang J. Shear wave elastography (SWE) is reliable method for testicular spermatogenesis evaluation after torsion. Int J Clin Exp Med. 2015 May 15;8(5):7089-97. eCollection 2015. PMID 26221246
- [Background] Kantarci F, Cebi Olgun D, Mihmanli I. Shear-wave elastography of segmental infarction of the testis. Korean J Radiol. 2012 Nov-Dec;13(6):820-2. doi: 10.3348/kjr.2012.13.6.820. Epub 2012 Oct 12. PMID 23118584
- [Background] Marcon J, Trottmann M, Rubenthaler J, Stief CG, Reiser MF, Clevert DA. Shear wave elastography of the testes in a healthy study collective - Differences in standard values between ARFI and VTIQ techniques. Clin Hemorheol Microcirc. 2016;64(4):721-728. doi: 10.3233/CH-168052. PMID 27935546
- [Background] Erdogan H, Durmaz MS, Ozbakir B, Cebeci H, Ozkan D, Gokmen IE. Experience of using shear wave elastography in evaluation of testicular stiffness in cases of male infertility. J Ultrasound. 2020 Dec;23(4):529-534. doi: 10.1007/s40477-020-00430-5. Epub 2020 Jan 30. PMID 31997228
- [Background] Yavuz A, Yokus A, Taken K, Batur A, Ozgokce M, Arslan H. Reliability of testicular stiffness quantification using shear wave elastography in predicting male fertility: a preliminary prospective study. Med Ultrason. 2018 May 2;20(2):141-147. doi: 10.11152/mu-1278. PMID 29730678
- [Background] Abdelaal AMA, El-Azizi HM, GamalEl Din SF, Abdulsalam Mohammad Azzazi O, Shokr Mohamed M. Evaluation of the potential role of shear wave elastography as a promising predictor of sperm retrieval in non-obstructive azoospermic patients: A prospective study. Andrology. 2021 Sep;9(5):1481-1489. doi: 10.1111/andr.13005. Epub 2021 Apr 25. PMID 33773055
- [Background] Rocher L, Criton A, Gennisson JL, Izard V, Ferlicot S, Tanter M, Benoit G, Bellin MF, Correas JM. Testicular Shear Wave Elastography in Normal and Infertile Men: A Prospective Study on 601 Patients. Ultrasound Med Biol. 2017 Apr;43(4):782-789. doi: 10.1016/j.ultrasmedbio.2016.11.016. Epub 2017 Jan 3. PMID 28062178
- [Background] Li M, Li FH, Du J, Wang ZQ, Zheng JF, Li Z, Ping P. [Quantitative analysis by real-time elastosonography for the differential diagnosis of azoospermia: preliminary application]. Zhonghua Nan Ke Xue. 2012 Jan;18(1):35-8. Chinese. PMID 22295846
- [Background] Hu JY, Huang WL, Gao Y, Yang Z, Ding L, Xie Y, Xie XY, Hu HT, Wang Z. Preliminary investigation of the diagnostic value of shear wave elastography in evaluating the testicular spermatogenic function in patients with azoospermia. Andrologia. 2021 Jun;53(5):e14039. doi: 10.1111/and.14039. Epub 2021 Mar 7. PMID 33682169
- [Background] Fu W, Cui J, Tang S. The relationship of testicular stiffness with Johnsen score and sperm retrieval outcome in men with non-obstructive azoospermia. Quant Imaging Med Surg. 2024 Apr 3;14(4):3033-3043. doi: 10.21037/qims-23-1381. Epub 2024 Mar 28. PMID 38617167
- [Background] Zhang H, Xi Q, Zhang X, Zhang H, Jiang Y, Liu R, Yu Y. Prediction of microdissection testicular sperm extraction outcome in men with idiopathic nonobstruction azoospermia. Medicine (Baltimore). 2020 May;99(18):e19934. doi: 10.1097/MD.0000000000019934. PMID 32358364
- [Background] Tunc L, Kirac M, Gurocak S, Yucel A, Kupeli B, Alkibay T, Bozkirli I. Can serum Inhibin B and FSH levels, testicular histology and volume predict the outcome of testicular sperm extraction in patients with non-obstructive azoospermia? Int Urol Nephrol. 2006;38(3-4):629-35. doi: 10.1007/s11255-006-0095-1. Epub 2006 Nov 3. PMID 17111079
- [Background] Amer M, Ateyah A, Zohdy W, Abd El Nasser T, Abdel-Malak G, Fakhry E. Preoperative and intraoperative factors that predict difficult testicular sperm retrieval in patients with nonobstructive azoospermia. Fertil Steril. 2002 Sep;78(3):646-7. doi: 10.1016/s0015-0282(02)03273-9. No abstract available. PMID 12215352